CLINICAL TRIAL: NCT01003080
Title: Unipolar vs. Bipolar Hemostasis in Total Knee Arthroplasty: A Prospective Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Sun Jin Kim, Chief of Adult Reconstruction, Montefiore Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 09-05-145
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Results first posted 2011-04-07 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Knee Arthroplasty
Keywords: The evaluation of hemostasis during total knee arthroplasty using the aquamantys device.

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- TKA with the Aquamantys for hemostasis (Experimental): This arm will receive the total knee arthroplasty with the Aquamantys device used for hemostasis.
  Interventions: Device: Aquamantys Device
- TKA without the Aquamantys for hemostasis (Active Comparator): This group will receive total knee arthroplasty using the standard treatment for hemostasis.
  Interventions: Other: Standard of care treatment for hemostasis during a total knee arthroplasty.

INTERVENTIONS:
Device: Aquamantys Device — The Aquamantys is used for hemostasis in patients randomized to receive total knee arthroplasty with the device.
  Arms: TKA with the Aquamantys for hemostasis
Other: Standard of care treatment for hemostasis during a total knee arthroplasty. — The active comparator arm will receive the "standard-of-care" for hemostasis during total knee arthroplasty. This is achieved with a unipolar Bovie electrocauterization device.
  Arms: TKA without the Aquamantys for hemostasis

SUMMARY:
The use of Aquamantys during total knee arthroplasty will reduce drain output and the necessity for blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Patient indicated for total knee arthroplasty

Exclusion Criteria:

* Patients undergoing revision total knee arthroplasty
* Patients with blood disorders
* Patients on chronic anti-thrombotic medication such as Coumadin
* Patients with a history of deep vein thrombosis
* Patients with a history of pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun Jin Kim, MD, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Jack D. Weiler Hospital-Division of Montefiore Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the medical clinics of Weiler and Montefiore hospitals under the Montefiore system in the Bronx, NY. Patients undergoing a total knee arthroplasty (TKA) were recruited over a 10 month period and either received hemostasis with the standard unipolar cauterizing device or the bipolar saline system.
Pre-assignment Details: Patients who were on anticoagulation therapy prior to their TKA were excluded from our study as this potentially would increase their amount of post-operative bleeding complicating the results of our study.
Period: Overall Study
Arm/Group | TKA With the Aquamantys for Hemostasis | TKA Without the Aquamantys for Hemostasis
Started | 50 | 61
Completed | 50 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TKA With the Aquamantys for Hemostasis | TKA Without the Aquamantys for Hemostasis | Total
Number analyzed (Participants) | 50 | 61 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 27 | 53
  >=65 years | 24 | 34 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (10.4) | 66.3 (9.6) | 66 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 51 | 89
  Male | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  United States | 50 | 61 | 111

OUTCOME MEASURES:

1. Primary Outcome: Drain Output.
Description: This is a measure of the average drain output collected in the first 24 hours following surgery.
Time Frame: First 24 hours following surgery.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | TKA With the Aquamantys for Hemostasis | TKA Without the Aquamantys for Hemostasis
Number analyzed (Participants) | 50 | 61
mL | 776 (334) | 778 (331.1)

ADVERSE EVENTS:
Arm/Group | TKA With the Aquamantys for Hemostasis | TKA Without the Aquamantys for Hemostasis
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/61
Other Adverse Events (participants affected / at risk) | 0/50 | 0/61

LIMITATIONS AND CAVEATS:
Operator dependent modifications may affect the standardization of the procedure; Surgeon is not blinded to the treatment used on each patient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No